CLINICAL TRIAL: NCT00807313
Title: Non-interventional Observational Study of Helical Tomotherapy for Oligometastatic Colorectal Cancer
Acronym: tomoligo
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Mark De Ridder, Head of Radiotherapy Department, Universitair Ziekenhuis Brussel
Other Study IDs: RCT501
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Colon Cancer; Rectal Cancer; Colorectal Cancer
Keywords: Oligometastatic disease; Colorectal cancer; Stereotactic body radiotherapy; Tomotherapy; Metabolic response; Stage IV
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- At best response: Patients with oligometastatic colorectal cancer, who presents at best response under chemotherapy, will receive stereotactic body radiotherapy on their residual disease
- No indication for chemotherapy: Patients with oligometastatic colorectal cancer, who are progressive under chemotherapy or who are no candidates for (further) chemotherapy, will receive stereotactic body radiotherapy on the sites of disease.

SUMMARY:
Patients with oligometastatic colorectal cancer (5 metastases or less) receive a combination of systemic treatment and often local treatment, such as surgery, radiofrequency ablation and more recently stereotactic body radiotherapy. The aim of this study is to register the results and side effects of stereotactic body radiotherapy (SBRT) by means of helical tomotherapy in the treatment of oligometastatic colorectal cancer.

The trial has two cohorts. Patients in cohort I get consolidation SBRT after best response on first line chemotherapy. Patients in cohort II get SBRT when there is progression under, or no indication for (further) chemotherapy. The primary endpoint is to evaluate the metabolic complete remission rate three months after the start of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with (residual) oligometastatic CRC: ≤ 5 mets
* Primary tumor treated with curative intention (surgery, radiotherapy, chemoradiotherapy)
* Functional liver volume > 1000cc if livermets, lung DLCO > 30% if lungmets.
* No Child B or C liver cirrhosis
* No contra-indications for radiation of all metastatic CRC (= no violation of constraints of organs at risk (OAR))
* No mets from another carcinoma
* Age > 18 years
* WHO-PS ≤ 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oligometastatic (5 metastases or less) colorectal cancer
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-12; Primary Completion 2011-07 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Metabolic complete remission rate | Three months

SECONDARY OUTCOMES:
Acute toxicity | Three months
Progression free survival | Three to thirty six months
Local control | Three to thirty six months
Survival | Three to thirty six months
Late toxicity | Three to thirty six months

CONTACTS AND LOCATIONS:
Overall Officials: Mark De Ridder, MD, PhD, Principal Investigator — UZ Brussel, Vrije Universiteit Brussel, dienst Radiotherapie
Locations (1):
- UZ Brussel, Vrije Universiteit Brussel, dienst Radiotherapie, Brussels, Belgium

REFERENCES:
- [Background] Verellen D, De Ridder M, Linthout N, Tournel K, Soete G, Storme G. Innovations in image-guided radiotherapy. Nat Rev Cancer. 2007 Dec;7(12):949-60. doi: 10.1038/nrc2288. PMID 18034185
- [Derived] Engels B, Gevaert T, Everaert H, De Coninck P, Sermeus A, Christian N, Storme G, Verellen D, De Ridder M. Phase II study of helical tomotherapy in the multidisciplinary treatment of oligometastatic colorectal cancer. Radiat Oncol. 2012 Mar 16;7:34. doi: 10.1186/1748-717X-7-34. PMID 22423615